CLINICAL TRIAL: NCT03845790
Title: Pharmacokinetic Study of Vancomycin, Clindamycin And/or Gentamicin Administration During Surgery Using a Microdialysis Procedure
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PK PROPHYLAXIE
Record Dates: First submitted 2019-02-15; First posted 2019-02-19 (Actual); Last update posted 2025-01-16 (Actual); Status verified 2025-01

CONDITIONS: Surgical Site Infection
MeSH Terms: conditions — Surgical Wound Infection | interventions — Blood Specimen Collection

STUDY DESIGN:
Intervention Model Description: Pharmacokinetic study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Blood and microdialysis samples — Blood and microdialisys pharmacocinetic samples on one of the two antibiotics prescribed in routine use

SUMMARY:
The surgical site infection is one of the most important causes of postoperative morbidity. The appropriate antibiotic prophylaxis is one of the most effective way to prevent surgical site infections. The beta-lactam are the most frequent antibiotics recommended for surgical prophylaxis and patients known to be allergic to beta-lactam are more likely to presented surgical site infection, probably due to use of others antibiotic such as vancomycin or clindamycin.

The main objective of the study is to describe the tissu and plasma pharmacokinetics of vancomycin, clindamycin and gentamicin using as surgical antibiotic prophylaxis in patients with beta-lactam hypersensivity and to predict the probability of target attainment for usual bacteria.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient between 18 and 80 years old
* Patient with history of beta-lactam hypersensitivity
* Patient who underwent abdominal or orthopedic surgery whose forseeable time exceeds 1 hour and requires a surgical antibiotic prophylaxis by vancomycin or clindamycin + gentamicin

Exclusion Criteria:

* morbid obesity (BMI > 35 kg/m2)
* mild to severe renal impairment (clearance creatinine < 60 ml/min)
* vancomycin, clindamycin or gentamicin hypersensitivity
* pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2019-05-26 (Actual); Primary Completion 2024-09-04 (Actual); Study Completion 2024-09-04 (Actual)

PRIMARY OUTCOMES:
Total and free plasma of vancomycin, clindamycin or gentamicin | 24 hours
Free tissue concentration of vancomycin, clindamycin or gentamicin every 20 minutes after the beginning of injections | 24 hours
Probability of target attainment of PK/PD index for usual bacteria (AUC/CMI >1 for vancomycin and clindamycin, Cmax/CMI >8 for gentamicin) with the recommended dosing regimen | 2 days

SECONDARY OUTCOMES:
Probability of target attainment of PK/PD index for usual bacteria (AUC/CMI >1 for vancomycin and clindamycin, Cmax/CMI >8 for gentamicin) with new simulated dosing regimens. | 2 days

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Poitiers, Poitiers, France

IPD SHARING:
Plan to Share IPD: No